CLINICAL TRIAL: NCT03661151
Title: Comparison of Treatment Effectiveness and Evaluation of Cost Between Surgical and Non-surgical Treatment for Gastroesophageal Reflux Disease (GERD)
Brief Title: Comparison of Treatment Outcome and Cost-effectiveness for GERD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sungsoo Park (Other)
Collaborators: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Kosin University Gospel Hospital (Other)
Responsible Party: Sponsor-Investigator, Sungsoo Park, Professor, Korea University Anam Hospital
Organization: Korea University Anam Hospital (Other)
Other Study IDs: GERD-PPI-ARS
Record Dates: First submitted 2018-06-15; First posted 2018-09-07 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal reflux disease; Antireflux surgery
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Antireflux surgery following PPI: A single cohort with the GERD patients who had acid suppressive medication with proton pump inhibitor (PPI) followed by laparoscopic antireflux surgery

SUMMARY:
This study was designed to evaluate the effectiveness of laparoscopic antireflux surgery for treatment of gastroesophageal reflux disease (GERD) comparing with that of non-surgical treatment.

DETAILED DESCRIPTION:
To treat GERD, the most patients with GERD are managed with acid suppressive medication first, and followed by antireflux surgery when the medical therapy is not effective or when the patient prefer surgery to quit the medicine.

This study has a single cohort in which the patient has the past history of GERD and medical treatment with proton pump inhibitors, and has scheduled to have laparoscopic antireflux surgery for treatment of GERD.

Treatment outcome of surgery will be evaluated comparing with the outcome of medical treatment before registration.

ELIGIBILITY:
Inclusion Criteria:

* Objectively diagnosed GERD
* Past history of medical treatment with PPI more than 8 weeks at any time before antireflux surgery
* Patients scheduled to undergo antireflux surgery to treat GERD

Exclusion Criteria:

* Other pathologic condition in upper gastrointestinal tract which needs surgical treatment
* No (or less than 8 weeks) past history of acid suppressive medical therapy with PPI
* Patients who underwent endoscopic antireflux procedure

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: GERD patients who have history of PPI therapy and scheduled to undergo antireflux surgery
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-02-25 (Actual); Primary Completion 2020-10-25 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptom Control Rate of Surgical and Non-surgical Treatment for Gastroesophageal Reflux Disease (GERD) | Change from baseline GERD symptom at 3 months after antireflux surgery
  GERD symptom control rate of surgical and non-surgical treatment for GERD based on the GERD symptom questionaire

SECONDARY OUTCOMES:
Medical Cost of Surgical and Non-surgical Treatment for Gastroesophageal Reflux Disease (GERD) | Change from baseline medical cost (non-surgical) at 3 months after antireflux surgery
  Evaluation of medical cost based on public insurance system and patients' history
Complication rate and adverse symptom rate related with antireflux surgery | Change from baseline GERD symptom at 3 months after antireflux surgery
  Surgical complication and adverse symptom related with antireflux surgery evaluated with GERD symptom questionaire and case records

CONTACTS AND LOCATIONS:
Overall Officials: Sungsoo Park, MD, PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea